CLINICAL TRIAL: NCT07326267
Title: Development and Evaluation of a School-Based Occupational Therapy Program Focused on Sensory Processing and Activities of Daily Living: A Randomized Controlled Trial
Brief Title: School-Based Sensory Processing and Daily Living Skills-Focused Occupational Therapy Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Feyza Şengül, Res. Asst., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2529c9d3ba6d4dce
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Intellectual Disability, Variable; Autism Spectrum Disorder (ASD)
Keywords: School-Based Occupational Therapy; Sensory Processing Intervention; Activities of Daily Living (ADL); Intellectual Disability (ID); Randomized Controlled Trial; Feasibility Trial; Goal Attainment Scaling (GAS); Special Education School; Independence; Sensory Integration
MeSH Terms: conditions — Intellectual Disability; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: After baseline assessment (T0), participants will be randomly allocated in a 1:1 ratio using concealed variable block randomization to either the intervention group or the active control group. The intervention group will receive a school-based occupational therapy program consisting of once-weekly 50-minute sessions over 10-12 weeks, including sensory preparation, task-oriented activities of daily living practice, and generalization. The active control group will receive family education, a written home program, and routine school monitoring.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- School-Based OT (Sensory + ADL) (Experimental): Participants receive a structured, school-based individual occupational therapy program targeting sensory processing and activities of daily living.
  Interventions: Behavioral: Individual School-Based Occupational Therapy Sessions; Behavioral: Sensory Preparation Using Proprioceptive, Vestibular, and Tactile Input; Behavioral: Task-Oriented Activities of Daily Living Training; Behavioral: Generalization and Classroom-Based Sensory Support Strategies; Behavioral: Family Education and Written Home Program
- Family Education and Home Program (Active Comparator): Participants receive family education and a written home program without individualized occupational therapy intervention.
  Interventions: Behavioral: Family Education and Written Home Program

INTERVENTIONS:
Behavioral: Individual School-Based Occupational Therapy Sessions — This intervention consists of individually delivered, school-based occupational therapy sessions conducted once weekly in 50-minute sessions over a period of 10-12 weeks. Sessions are implemented in a designated therapy space within the school environment and are guided by a predefined intervention protocol to ensure standardization while allowing individualization based on each child's needs.
  Each session is planned and delivered by a trained occupational therapist and targets functional participation within daily school routines. Intervention content is individualized according to the child's sensory processing profile, functional performance, and prioritized activities of daily living goals. Session fidelity is monitored using structured checklists to ensure adherence to the protocol across the intervention period.
  Other Names: Intervention 1
  Arms: School-Based OT (Sensory + ADL)
Behavioral: Sensory Preparation Using Proprioceptive, Vestibular, and Tactile Input — IThis intervention component involves structured sensory preparation activities implemented at the beginning of each individual occupational therapy session. Sensory preparation is designed to support arousal regulation, attention, and readiness for task engagement by providing individualized proprioceptive, vestibular, and tactile input.
  Sensory strategies are selected based on each child's sensory processing characteristics and observed regulation needs and may include activities such as deep pressure input, controlled movement experiences, and tactile modulation tasks. The intensity, duration, and combination of sensory inputs are adjusted within a standardized framework to optimize engagement in subsequent task-oriented activities.
  Other Names: Intervention 2
  Arms: School-Based OT (Sensory + ADL)
Behavioral: Task-Oriented Activities of Daily Living Training — This intervention component focuses on task-oriented training targeting individualized activities of daily living relevant to the child's school and daily life contexts. Activities are selected collaboratively based on assessment findings and may include self-care and school-related daily living tasks such as hand washing, eating, dressing, organizing personal belongings, and waiting in line.
  Training emphasizes active participation, graded task demands, and repeated practice within meaningful contexts. Tasks are adapted to the child's current performance level to promote skill acquisition, independence, and functional efficiency. Performance is supported through appropriate cueing, environmental modification, and adaptive strategies as needed. Progress toward individualized goals is monitored throughout the intervention period and informs ongoing task selection and grading.
  Other Names: Intervention 3
  Arms: School-Based OT (Sensory + ADL)
Behavioral: Generalization and Classroom-Based Sensory Support Strategies — This intervention component focuses on supporting the generalization and sustainability of gains achieved during individual occupatinal therapy sessions by embedding sensory and task-related strategies into natural school and home contexts. Structured generalization activities are implemented to facilitate the transfer of individualized activities of daily living skills from therapy sessions to classroom routines and daily life environments.
  As part of this component, brief classroom-based sensory support strategies ("sensory micro-protocols") are introduced through teacher guidance. These strategies are designed to promote sensory regulation and participation during typical classroom activities (e.g., transitions, seated tasks, waiting periods) without disrupting routine educational flow. Teachers are provided with clear, feasible guidance on when and how to apply these strategies in response to children's sensory regulation needs.
  Other Names: Intervention 4
  Arms: School-Based OT (Sensory + ADL)
Behavioral: Family Education and Written Home Program — This intervention consists of structured family education and a written home program focused on supporting children's activities of daily living within the home environment. Families receive guidance on daily living routines, environmental organization, and basic strategies to support independence and participation in everyday tasks. Educational content is provided in a standardized written format to ensure consistency across participants.
  No individualized occupational therapy sessions or direct therapeutic intervention are delivered to participants in this group during the study period. Children continue their routine school activities and standard school monitoring.
  Other Names: Intervention 5

SUMMARY:
This study aims to develop and evaluate a school-based occupational therapy program focused on sensory processing and activities of daily living for children with Autism Spectrum Disorder and Intellectual Disability. Sensory processing difficulties often affect school participation, behavior regulation, and independence in daily tasks. Although occupational therapy interventions have shown benefits in clinical settings, evidence for their use in schools is limited.

The trial will take place at Vali Ayhan Çevik Special Education School and will enroll students aged 6 to 14 years. Participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive weekly 50-minute occupational therapy sessions for 10 to 12 weeks, including sensory preparation, task-oriented practice, and strategies to support everyday skills. The control group will receive family education, a written home program, and routine school observation.

Outcomes will be assessed at baseline, after the intervention, and at 4 to 6-week follow-up. The main outcome is change in Goal Attainment Scaling scores, which reflect progress toward individualized goals. Additional measures include functional ability, sensory processing, and demographic and clinical information. The study will also monitor feasibility and how closely the program is delivered as planned.

This research is expected to provide evidence on the feasibility and effects of a standardized occupational therapy program in a school setting and to support the use of similar approaches in educational contexts.

DETAILED DESCRIPTION:
This project aims to develop and evaluate a School-Based Occupational Therapy Program focused on Sensory Processing and Activities of Daily Living (ADL) through a randomized controlled feasibility trial. Children with Autism Spectrum Disorder (ASD) and Intellectual Disability (ID) frequently experience sensory processing difficulties that adversely affect school participation, behavioral regulation, and independence in ADLs. Although the effectiveness of sensory-based and ADL-focused occupational therapy interventions has been demonstrated in clinical settings, evidence regarding their standardized, high-fidelity implementation within school environments remains limited.

The study will be conducted at Vali Ayhan Çevik Special Education School and will include students aged 6-14 years. Using a two-arm, parallel-group randomized controlled design, participants will be randomly allocated (1:1) to either an intervention group or a control group. The intervention group will receive once-weekly, 50-minute occupational therapy sessions over 10-12 weeks, comprising sensory preparation, task-oriented ADL practice, and generalization activities. The control group will receive family education, a written home program, and routine school observation. Outcome assessments will be conducted at baseline (T0), post-intervention (T1), and follow-up (T2; 4-6 weeks).

The primary outcome measure will be the Goal Attainment Scaling (GAS) T-score, reflecting progress toward individualized, occupation-based goals. Secondary outcomes will include the Pediatric Disability Assessment Inventory (PEDI), Sensory Profile, and a Pediatric Information Form capturing demographic and clinical routine data. Feasibility indicators-such as attendance rate, data completeness, and classroom micro-protocol utilization-as well as intervention fidelity measures, including session checklists and secondary rater/video-based evaluations, will be systematically monitored.

Expected outcomes include clinically meaningful improvements in GAS scores and ADL-related indicators in the intervention group, alongside enhanced sensory equipment infrastructure and the development of teacher micro-protocols to strengthen institutional capacity. This study aims to address a significant gap in the literature on school-based occupational therapy in Türkiye by providing a feasible, standardized, and replicable intervention model for special education settings.

ELIGIBILITY:
Inclusion Criteria:

* Regular school attendance (Anticipated ability to attend at least 70% of the planned intervention sessions during the study period);
* Written informed consent obtained from the family;
* Formal diagnosis of Autism Spectrum Disorder or Intellectual Disability, documented by an official disability report;
* Presence of observable difficulties in sensory processing and activities of daily living (ADL), verified through the student's Individualized Education Program (IEP) records;
* Ability to partially follow single-step basic instructions, as documented in the IEP records;
* Willingness of families and teachers to participate in follow-up assessments (T2 and beyond).

Exclusion Criteria:

* Uncontrolled epilepsy or other medical conditions that may interfere with participation or safety during sessions.
* Medical contraindications to modalities such as swinging or deep pressure or severe musculoskeletal limitations preventing participation in task-oriented ADL practice.
* Being in a period of severe acute behavioral crisis;
* Concurrent participation in occupational therapy or special education programs for ≥2 hours per week that would compromise data interpretation;
* Presence of severe visual or hearing impairments that would substantially limit the child's ability to perceive sensory stimuli, follow task instructions, or validly engage in assessment procedures;
* Inability to maintain family and/or teacher collaboration throughout the intervention period;
* Inconsistent school attendance during the intervention period (e.g., prolonged absenteeism);
* Insufficient language comprehension to engage with basic task instructions even with support.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scaling | Baseline (T0), post-intervention at 10-12 weeks (T1), and follow-up at 4-6 weeks after the intervention (T2)
  It is a method developed to measure progress toward individualized goals and provides a sensitive way to monitor clinical change, particularly in populations with heterogeneous profiles and in contexts relying on subjective outcome measures. Originally developed by Kiresuk and Sherman, Goal Attainment Scaling (GAS) evaluates goal achievement using a five-point scale ranging from -2 (much less than the expected outcome) to +2 (much more than the expected outcome), with 0 representing the expected level of performance. The scale is based on measurable and behaviorally defined goals collaboratively established by the individual, family, and therapist. Each goal can be weighted according to its importance and level of difficulty (weight = importance × difficulty).Recent studies have highlighted GAS as a sensitive, clinically meaningful, and participant-centered outcome measure in pediatric rehabilitation and occupational therapy practice.

SECONDARY OUTCOMES:
Sensory Profile | Baseline (T0), post-intervention at 10-12 weeks (T1), and follow-up at 4-6 weeks after the intervention (T2)
  Sensory Profile is an assessment tool developed by occupational therapist Winnie Dunn to evaluate sensory processing characteristics in children. It was designed for use with children aged 3-10 years and assesses children's responses to sensory stimuli during daily life activities based on caregiver observations. The scale consists of 125 items and is completed by the caregiver in approximately 30-40 minutes. Each item is rated on a 5-point Likert scale-"Always," "Frequently," "Occasionally," "Seldom," and "Never"-with scores ranging from 1 (Always) to 5 (Never). Lower scores indicate more pronounced sensory processing difficulties. The scale is organized into three main sections-sensory processing, modulation, and behavioral-emotional responses-and includes 14 derived subfactors. The Turkish version has demonstrated acceptable to high internal consistency. Although the normative age range of the test is 3-10 years, its use with children up to 14 years of age has also been reported
Pediatric Evaluation of Disability Inventory (PEDI) | Baseline (T0), post-intervention at 10-12 weeks (T1), and follow-up at 4-6 weeks after the intervention (T2)
  It was developed by Haley et al. to assess functional skills and performance levels in children. Although it was originally designed for children aged 6 months to 7.5 years, it can also be used with older children who show limitations in functional performance. The scale consists of three main components-functional skills, caregiver assistance, and modifications-each covering the domains of self-care, mobility, and social function. The functional skills component evaluates the child's level of independence using a "capable/incapable" rating, while the caregiver assistance component is scored on a scale ranging from 0 (total dependence) to 5 (independence).

OTHER OUTCOMES:
Pediatric Information Form | Baseline (T0)
  The Pediatric Information Form is a structured data collection tool used to comprehensively assess children's developmental, sensory, motor, language, self-care, and social skills. It systematically gathers information on the child's demographic characteristics, medical and developmental history, parental observations, therapy background, and daily living routines. In this study, the form will be used as a pre-intervention assessment to support a holistic characterization of participants' sensory processing and daily living skills profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyhun Türkmen, associate professor, Principal Investigator — Çankırı Karatekin University, Faculty of Health Sciences, Department of Occupational Therapy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions, data protection regulations, and the involvement of a pediatric population in a school-based setting.

REFERENCES:
- [Background] Schaaf RC, Burke JP, Cohn E, May-Benson TA, Schoen SA, Roley SS, Lane SJ, Parham LD, Mailloux Z. State of measurement in occupational therapy using sensory integration. Am J Occup Ther. 2014 Sep-Oct;68(5):e149-53. doi: 10.5014/ajot.2014.012526. PMID 25184475
- [Background] Haley SM. Pediatric Evaluation of Disability Inventory (PEDI): Development, standardization and administration manual. (No Title). 1992.
- [Background] Mailloux Z, May-Benson TA, Summers CA, Miller LJ, Brett-Green B, Burke JP, Cohn ES, Koomar JA, Parham LD, Roley SS, Schaaf RC, Schoen SA. Goal attainment scaling as a measure of meaningful outcomes for children with sensory integration disorders. Am J Occup Ther. 2007 Mar-Apr;61(2):254-9. doi: 10.5014/ajot.61.2.254. PMID 17436848
- [Background] Kiresuk TJ, Sherman RE. Goal attainment scaling: A general method for evaluating comprehensive community mental health programs. Community Ment Health J. 1968 Dec;4(6):443-53. doi: 10.1007/BF01530764. PMID 24185570
- [Background] Laverdure P, Beisbier S. Occupation- and Activity-Based Interventions to Improve Performance of Activities of Daily Living, Play, and Leisure for Children and Youth Ages 5 to 21: A Systematic Review. Am J Occup Ther. 2021 Jan-Feb;75(1):7501205050p1-7501205050p24. doi: 10.5014/ajot.2021.039560. PMID 33399053
- [Background] Grandisson M, Rajotte E, Godin J, Chretien-Vincent M, Milot E, Desmarais C. Autism spectrum disorder: How can occupational therapists support schools? Can J Occup Ther. 2020 Feb;87(1):30-41. doi: 10.1177/0008417419838904. Epub 2019 Aug 11. PMID 31401850
- [Background] Ouellet B, Carreau E, Dion V, Rouat A, Tremblay E, Voisin JIA. Efficacy of Sensory Interventions on School Participation of Children With Sensory Disorders: A Systematic Review. Am J Lifestyle Med. 2018 Jul 11;15(1):75-83. doi: 10.1177/1559827618784274. eCollection 2021 Jan-Feb. PMID 33447172
- [Background] Lynch H, Moore A, O'Connor D, Boyle B. Evidence for Implementing Tiered Approaches in School-Based Occupational Therapy in Elementary Schools: A Scoping Review. Am J Occup Ther. 2023 Jan 1;77(1):7701205110. doi: 10.5014/ajot.2023.050027. PMID 36706276
- [Background] Cahill S, Bazyk S. School-based occupational therapy. Case-Smith's occupational therapy for children and adolescents. 2020:627-58.
- [Background] Jeong EH. Effects of school-based occupational therapy program for children with disabilities in elementary school in Korea: a case study. BMC Psychol. 2024 Jan 16;12(1):26. doi: 10.1186/s40359-024-01520-3. PMID 38229207